CLINICAL TRIAL: NCT07152275
Title: The Effect of Percussive Therapy on Muscle Flexibility, Balance, and Jump Performance in Licensed U19 Football Players and Sedentary Healthy Males Under 19 Years of Age
Brief Title: Percussive Therapy in U19 Males: Flexibility, Balance, Jump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Percussive Therapy
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Physical Inactivity; Postural Balance; Athletic Performance
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Non-Randomized, Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Licensed U19 Football Players) (Experimental): This group includes male adolescents aged 15-19 who have an active football license and engage in regular sports activity.
  Intervention:
  Name: Percussive Therapy Description: A 120-second percussive therapy protocol will be applied to each participant's hamstring muscles using a handheld massage gun (Hypervolt Go 2). The treatment includes 60 seconds on the semitendinosus and semimembranosus, and 60 seconds on the biceps femoris, performed while the participant is in a prone position.
  Timing: Single session Device Used: Hypervolt Go 2 massage gun
  Interventions: Device: Percussive Therapy
- Sedentary Group (Non-Athlete Healthy Males) (Experimental): This group includes healthy male adolescents aged 15-19 who have not engaged in regular physical activity in the past 6 months and have a BMI below 25.
  Intervention:
  Name: Percussive Therapy Description: The same 120-second percussive therapy protocol will be applied as in the active group, under identical conditions and using the same device.
  Timing: Single session Device Used: Hypervolt Go 2 massage gun
  Interventions: Device: Percussive Therapy

INTERVENTIONS:
Device: Percussive Therapy — Percussive therapy will be administered using the "Hypervolt Go 2 Black," a massage gun commonly used in clinical and athletic settings.
  Participants will lie in a prone position on a treatment table. To promote hamstring muscle relaxation, a support roll will be placed under the ankle. The intervention will be delivered by the same researcher for all participants to ensure consistency. Using the round head attachment, percussive therapy will be applied longitudinally along the hamstring muscle group (from proximal to distal) for a total of 120 seconds per leg. Specifically, 60 seconds will be applied to the semitendinosus and semimembranosus, and 60 seconds to the biceps femoris. The same procedure will then be repeated on the opposite leg.

SUMMARY:
This study aims to evaluate the effects of percussive therapy on muscle flexibility, balance, and jump performance in licensed U19 football players and sedentary healthy males under 19. Percussive therapy will be applied to the hamstring muscles for 120 seconds. Flexibility, balance, and explosive strength will be assessed using the sit-and-reach test, Y-Balance Test, and vertical jump test, respectively. The study also aims to compare the therapy's effects between active and sedentary participants.

DETAILED DESCRIPTION:
This study investigates the effects of 120-second percussive therapy applied to the hamstring muscles on flexibility, balance, and jump performance in two distinct groups: licensed U19 football players and sedentary healthy males under the age of 19. The intervention will be delivered using a handheld massage gun device, and outcomes will be evaluated using the sit-and-reach test (flexibility), the Y-Balance Test (dynamic balance), and the My Jump Lab mobile app (jump performance). Pre- and post-intervention assessments will be compared within each group, and the results will also be analyzed to identify any differences in response between the active and sedentary participants.

ELIGIBILITY:
Inclusion Criteria: (Participants must meet all of the following to be eligible.)

* Male individuals aged 15 to 19 years
* Voluntarily agreeing to participate

  **For the athlete group:
* Actively licensed U19 football player

  **For the sedentary group:
* No regular physical activity for the past 6 months
* Body Mass Index (BMI) under 25 kg/m2
* Physical activity level below 3000 MET-min/week as assessed by the International Physical Activity Questionnaire (IPAQ)

Exclusion Criteria: (Participants will be excluded if they meet any of the following.)

* Presence of acute or chronic lower extremity injuries
* History of lower extremity surgery
* Inability to tolerate percussive therapy
* Leg length discrepancy
* Restricted lower extremity joint range of motion due to any condition

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Change in Hamstring Flexibility | Within 1 hour (pre- and post-intervention)
  Flexibility will be assessed using the sit-and-reach test before and after percussive therapy. The best of three attempts (in centimeters) will be recorded.
Change in Dynamic Balance | Within 1 hour (pre- and post-intervention)
  Balance will be evaluated using the Y-Balance Test in three directions (anterior, posteromedial, and posterolateral). Results will be normalized based on leg length and averaged (% of leg length).
Change in Vertical Jump Performance | Within 1 hour (pre- and post-intervention)
  Explosive strength will be measured using the My Jump Lab app, which calculates jump height and flight time. The best result of the three trials (in centimeters) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Batuhan Kaykusuz, Principal Investigator — Yuksek Ihtisas University; Rashıd Karımzade, Principal Investigator — Yuksek Ihtisas University; Busra Kalkan Balak, Study Director — Yuksek Ihtisas University; Gungor Beyza Ozvar Senoz, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No